CLINICAL TRIAL: NCT06673784
Title: Evaluation and Risk Factors of Post-traumatic Endophthalmitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer Gamal AbdElmohsen Ahmed, Doctor, Assiut University
Other Study IDs: Ev. of post-traumatic Endoph.
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis | interventions — Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Evaluation of post-traumatic endophthalmitis: 1. conception
  2. acquisition of data
  3. analysis of data
  Interventions: Diagnostic Test: ophthalmic saline eye drops; Drug: Saline

INTERVENTIONS:
Diagnostic Test: ophthalmic saline eye drops — for optical examination
Drug: Saline — Most one natural and not effects on study

SUMMARY:
1. identify the incidence of post-traumatic endophthalmitis and the related risk factors influencing its development.
2. study the clinical- microbiological profile and evaluate the functional and anatomical outcomes of post-traumatic endophthalmitis (PPTE).

ELIGIBILITY:
Inclusion Criteria:

* Patients exposed to eye trauma and developed post-traumatic endophthalmitis

Exclusion Criteria:

* Patients who refuse to sign informed consent in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Evaluation and risk factors of post-traumatic endophthalmitis with general and optical examination on patients exposed to eye trauma and developed post-traumatic endophthalmitis
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Knowledge of clinical features outcomes of post-traumatic endophthalmitis | Baseline
  Knowledge of clinical features which will be shown due to post-traumatic endophthalmitis

SECONDARY OUTCOMES:
The factors associated with a worse prognosis in post-traumatic endophthalmitis | Baseline
  Discrimination the worst prognosis in post-traumatic endophthalmitis

REFERENCES:
- [Background] Alfaro DV, Roth DB, Laughlin RM, Goyal M, Liggett PE. Paediatric post-traumatic endophthalmitis. Br J Ophthalmol. 1995 Oct;79(10):888-91. doi: 10.1136/bjo.79.10.888. PMID 7488575